CLINICAL TRIAL: NCT03647241
Title: An Evaluation of the Efficacy of Self-Ligating Brackets Alone Or In Combination With Flapless Corticotomy In Leveling And Aligning Severely Crowded Dental Arches Compared With Conventional Brackets: A Randomized Clinical Controlled Trial
Brief Title: Evaluation of Self-ligating Brackets Plus Minor Surgery in Treating Crowded Cases of Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-10-2018
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Malocclusion of Anterior Teeth
MeSH Terms: interventions — Piezosurgery; Cerebral Decortication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Ligating Brackets (Experimental): Patients will be treated using self-ligating brackets to achieve proper alignment of teeth
  Interventions: Device: Self-Ligating Brackets
- Self-Ligating Brackets with Corticotomy (Experimental): Patients will be treated using self-ligating brackets with corticotomy (alveolar cortical cuts) in order to accelerate orthodontic treatment.
  Interventions: Device: Self-Ligating Brackets; Procedure: Corticotomy
- Traditionally-Ligated Brackets (Active Comparator): Patients in this group will be treated using traditionally-ligated brackets to achieve proper alignment of teeth
  Interventions: Device: Traditionally-Ligated Brackets

INTERVENTIONS:
Device: Self-Ligating Brackets — These brackets can be opened and closed through the use of a sliding cap embedded into the design of these brackets. There is no need to use elastic modules to ligate the arch.
  Other Names: SLBs
  Arms: Self-Ligating Brackets; Self-Ligating Brackets with Corticotomy
Device: Traditionally-Ligated Brackets — These brackets are used in the conventional manner, where the orthodontist is obliged to use elastic modules to engage the arch into the slot of the bracket.
  Other Names: Non-SLBs
  Arms: Traditionally-Ligated Brackets
Procedure: Corticotomy — Corticotomy without flap elevations will be performed in order to induce acceleration in tooth movement during the orthodontic treatment in only one group.
  Other Names: Piezosurgery; Decortication
  Arms: Self-Ligating Brackets with Corticotomy

SUMMARY:
Patients at the Orthodontic Department of University of Damascus Dental School will be examined and subjects who meet the inclusion criteria will be admitted then the initial diagnostic records (diagnostic gypsum samples - internal and external oral photographs as well as radiographic images) will be studied to ensure that the selection criteria are accurately matched.

The aim of this study is to compare three groups of patients with severe crowding of the upper anterior teeth:

* Group 1 : Patients will be treated using self-ligating brackets
* Group 2 : Patients will be treated using self-ligating brackets associated with flapless corticotomy.
* Group 3 : Patients will be treated using traditional brackets (i.e. brackets positioned on the labial surface of the teeth)

At the end of leveling and aligning phase, we will compare the self-ligating brackets and traditional brackets ( the acceleration of teeth movement, dental and alveolar changes and other variables ) Also, there is an intention to study the effectiveness of using flapless corticotomy with the self-ligating brackets.

DETAILED DESCRIPTION:
The sample of this study will be chosen according the following steps:

* The examination of patients referred to the Department of Orthodontics at the University of Damascus Dental School (clinical examination, diagnostic plaster models, radiographic photos , external and internal oral photographs) then subjects who meet the inclusion criteria will be included in this trial.
* A random sample of 100 patients from the sampling frame will be chosen.
* An information sheet ( including the research objective and treatment plan in detail ) will be given to each candidate. Then consent forms will be collected from those who agree to participate.
* A random selection of 60 patients will be performed. Then a random distribution of these patients to 3 groups will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients: 17-28 years.
2. Severe crowding greater than 6 mm on the upper jaw in which orthodontic treatment requires at least two upper extraction.
3. The Little's Index of Irregularity is over 7 mm.
4. There is no previous orthodontic treatment.
5. The patient dose not take any drug may interfere with the tooth movement (Cortisone, NSAIDs, ...).
6. The patient has good oral health (i.e., Plaque Index is less or equal to 1 according to Loe and Silness (1963).
7. Class I or mild class II (ANB ≤ 5) or mild class III (ANB ≥ 0) skeletal relationship.
8. Overbite is between 0-4 mm.
9. There is no skeletal constriction on the upper jaw.
10. Full presence of all permanent teeth in the dental arch (except for third molars)

Exclusion Criteria:

1. Any systemic diseases that would affect tooth movement .
2. Any congenital syndromes or cleft lip and palate cases
3. Bad oral health

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Duration of Alignment | This variable is going to be measured at the end of the alignment stage (i.e. expected to occur within four to six months)
  The time required in days will be calculated from the beginning of treatment till the end of the alignment stage
Change in Little's Index | T0: one day before the beginning of treatment; T1: after one month; T2: after two months; T3: after three months; T4: after four months; T5: at the end of the alignment stage (which is expected to occur within 4 to 6 months)
  The irregularity of the upper and lower incisors is calculated by measuring the amount of deviation of the anatomic contact points between the six incisors in the horizontal direction in mm, since the sum of these measurements represents the value of the index (Little, 1975). The more the score is, the more crowded the case is.
Change in inter-canine width lingually | T1: One day before the beginning of treatment; T2: at the end of the alignment stage (is expected within four to six months)
  The distance between the most lingual points on the lingual surface of the canines on the upper dental arch. This will be measured on plaster models.
Change in inter-canine width | T1: One day before the beginning of treatment; T2: at the end of the alignment stage (is expected within four to six months)
  The distance between the cusp tips of the upper canines. This variable will be measured on plaster models.
Change in Canine Rotation Angle | T1: One day before the beginning of treatment; T2: at the end of the alignment stage (is expected within four to six months)
  It is calculated by the angle formed between the median palatine suture and the line passing through the two medial and lateral contact points of the canine.
Change in Lateral Incisor Rotation Angle | T1: One day before the beginning of treatment; T2: at the end of the alignment stage (is expected within four to six months)
  It is calculated by the angle formed between the median palatine suture and the line passing through the two medial and lateral contact points of the lateral incisor.
Change in Central Incisor Rotation Angle | T1: One day before the beginning of treatment; T2: at the end of the alignment stage (is expected within four to six months)
  It is calculated by the angle formed between the median palatine suture and the line passing through the two medial and lateral contact points of the central incisor.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Al-Ibrahim, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Issam Khoury, DDS MSc PhD, Study Director — Professor of Oral and Maxillofacial Surgery, Oral and Maxillofacial Surgery Department, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang X, Xue C, He Y, Zhao M, Luo M, Wang P, Bai D. Transversal changes, space closure, and efficiency of conventional and self-ligating appliances : A quantitative systematic review. J Orofac Orthop. 2018 Jan;79(1):1-10. doi: 10.1007/s00056-017-0110-4. Epub 2017 Nov 3. PMID 29101414
- [Background] Yang X, Su N, Shi Z, Xiang Z, He Y, Han X, Bai D. Effects of self-ligating brackets on oral hygiene and discomfort: a systematic review and meta-analysis of randomized controlled clinical trials. Int J Dent Hyg. 2017 Feb;15(1):16-22. doi: 10.1111/idh.12220. Epub 2016 Apr 20. PMID 27095145
- [Background] Yang X, He Y, Chen T, Zhao M, Yan Y, Wang H, Bai D. Differences between active and passive self-ligating brackets for orthodontic treatment : Systematic review and meta-analysis based on randomized clinical trials. J Orofac Orthop. 2017 Mar;78(2):121-128. doi: 10.1007/s00056-016-0059-8. Epub 2017 Feb 21. PMID 28224175
- [Background] Qamruddin I, Alam MK, Mahroof V, Fida M, Khamis MF, Husein A. Effects of low-level laser irradiation on the rate of orthodontic tooth movement and associated pain with self-ligating brackets. Am J Orthod Dentofacial Orthop. 2017 Nov;152(5):622-630. doi: 10.1016/j.ajodo.2017.03.023. PMID 29103440
- [Background] Nahas AZ, Samara SA, Rastegar-Lari TA. Decrowding of lower anterior segment with and without photobiomodulation: a single center, randomized clinical trial. Lasers Med Sci. 2017 Jan;32(1):129-135. doi: 10.1007/s10103-016-2094-5. Epub 2016 Oct 20. PMID 27761668
- [Background] Hassan SE, Hajeer MY, Alali OH, Kaddah AS. The Effect of Using Self-ligating Brackets on Maxillary Canine Retraction: A Split-mouth Design Randomized Controlled Trial. J Contemp Dent Pract. 2016 Jun 1;17(6):496-503. doi: 10.5005/jp-journals-10024-1879. PMID 27484605
- [Background] Charavet C, Lecloux G, Bruwier A, Rompen E, Maes N, Limme M, Lambert F. Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res. 2016 Aug;95(9):1003-9. doi: 10.1177/0022034516645066. Epub 2016 Apr 29. PMID 27129491
- [Background] Wahab RM, Idris H, Yacob H, Ariffin SH. Comparison of self- and conventional-ligating brackets in the alignment stage. Eur J Orthod. 2012 Apr;34(2):176-81. doi: 10.1093/ejo/cjq179. Epub 2011 Apr 8. PMID 21478298
- [Background] Scott P, DiBiase AT, Sherriff M, Cobourne MT. Alignment efficiency of Damon3 self-ligating and conventional orthodontic bracket systems: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2008 Oct;134(4):470.e1-8. doi: 10.1016/j.ajodo.2008.04.018. PMID 18929262